CLINICAL TRIAL: NCT01888640
Title: Fibromyalgia Activity Study With Transcutaneous Electrical Nerve Stimulation
Brief Title: Fibromyalgia Activity Study With Transcutaneous Electrical Nerve Stimulation (FAST)
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen Sluka (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor-Investigator, Kathleen Sluka, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201110717
Record Dates: First submitted 2013-06-13; First posted 2013-06-28 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia
Keywords: TENS; Fibromyalgia; Accelerometer
MeSH Terms: conditions — Fibromyalgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- ActiveTENS (Active Comparator): Active TENS for 4 weeks of the study and will add an additional 4 weeks of active TENS for the last 4 weeks of the study.
  Interventions: Device: TENS
- Placebo TENS (Placebo Comparator): This group will receive placebo TENS for the first 4 weeks of the study and then active TENS for the last four weeks of the study.
  Interventions: Device: TENS
- No TENS (Standard Care) (No Intervention): Participants will not receive TENS intervention during the first 4 weeks of the trial but will complete all testing procedures as the other two arms. This group will receive active TENS during the last 4 weeks of the study.

INTERVENTIONS:
Device: TENS — TENS Parameters: Active TENS and Placebo TENS
  * TENS Frequency - 2-125 Hz
  * TENS Pulse Width - 200 µs
  * TENS Intensity - Maximal tolerable intensity
  * Duration: 2 hours per day. The 2 hours may be broken into smaller segments of time with a minimum of 30 minutes.
  * Administration - Daily
  * TENS Location: TENS electrode on the skin will be a 4 x 7 butterfly electrode to the cervical and lumbar region.
  Placebo TENS Unit Active TENS unit No TENS - Standard Care
  Other Names: Empi Select Unit
  Arms: ActiveTENS; Placebo TENS

SUMMARY:
Pain associated with fibromyalgia interferes with daily function, work, and social activities resulting in a decreased quality of life. People with fibromyalgia also have a significant amount of fatigue and a fear of movement. People with fibromyalgia show enhanced excitability of pain neurons in the central nervous system and reduced pain inhibition. Therefore, one of the main treatments for patients with fibromyalgia must focus on pain relief to allow the person to function more independently both at home and at work. Transcutaneous electrical nerve stimulation is used by health professionals to deliver electrical stimulation through the skin for pain control. Basic science studies, from the PI's laboratory show that TENS activates descending pain inhibitory pathways to inhibit excitability of pain neurons. Thus the ideal patient population for the treatment of TENS would be one in which there is enhanced central excitability and reduced inhibition; fibromyalgia is such a condition.

Hypothesis: The investigators hypothesize that application of Transcutaneous Electrical Nerve Stimulation (TENS) to patients with fibromyalgia will reduce resting and movement-related pain and reduce central excitability by restoring diffuse noxious inhibitory controls (DNIC), and that this decrease in pain and/or central excitability will reduce fatigue and fear of movement, thereby improving function and quality of life

DETAILED DESCRIPTION:
This is a phase II randomized, double-blind, placebo controlled multi-center clinical trial involving a device, Transcutaneous Electrical Nerve Stimulation (TENS). TENS is a non-pharmacological agent which delivers electrical stimulation by a battery operated device via electrodes placed on the skin. TENS is considered to be a safe, inexpensive and non-invasive modality used to treat a variety of acute and chronic pain conditions. The initial phase of the study will randomly allocate subjects to receive active TENS, placebo TENS or standard care (No TENS). After participating in the 1 month random assignment, all subjects will receive active TENS for 1 month. The subjects will make 4 visits to the clinic approximately 2 to 3 1/2 hours each visit. Visits will entail questionnaires, functional tasks, accelerometry, TENS, pain and fatigue assessments.

Study Aims:

Aim #1: The primary aim of the study is to test the effectiveness of repeated TENS use on movement-related pain in people with fibromyalgia with random assignment to three treatments: standard care, placebo TENS and active Aim #2: A secondary aim will test if pain reduction by TENs results in a concomitant decrease in fatigue and fear of movement, and an increase in function and quality of life. Outcome measures will include physical function by directly assessing daily activity with an accelerometer, as well as performing specific functional tasks

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18 to 70 years of age
* Women may participate in the study, with the understanding that within the clinical population of fibromyalgia the there is a 7:1 ratio of female to male.
* Diagnosis of Fibromyalgia by 1990 ACR criteria (11/18 tender points)
* History of cervical or lumbar pain with fibromyalgia (this is expected in all patients since axial pain is required for diagnosis)
* Current stable treatment regimen for the last 4 weeks and projected stable treatment regimen for the next 2 months.
* English speaking

Exclusion Criteria:

* Current or history of cardiovascular, pulmonary, neurological, endocrine, or renal disease that would preclude the involvement in the study.
* TENS use in the last 5 years
* Pacemaker
* Uncontrolled blood pressure or diabetes
* Neuropathic pain condition
* Systemic autoimmune disorder (Lupus, PMR, RA, Psoriasis, Psoriatic arthritis)
* Spinal fusion - cervical or lumbar
* Metal implants in cervical or lumbar region
* Severe skin allergy to adhesive
* Allergy to nickel
* Pain level less than 4
* Pregnancy
* Epilepsy
* Change in or new drug or treatment program within the last month or in the next 2months, i.e. must have a stable treatment plan
* Unstable medical or psychiatric condition which in the opinion of the investigator could compromise the subject's welfare or confound the study results

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Sluka, PhD, PT, Principal Investigator — University of Iowa; Leslie J. Crofford, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
By publication
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available by publication by April 2019 and for one year after closeout of the study and upon request with a proposed study protocol for 5 years.

REFERENCES:
- [Background] Sluka KA, Vance CG, Lisi TL. High-frequency, but not low-frequency, transcutaneous electrical nerve stimulation reduces aspartate and glutamate release in the spinal cord dorsal horn. J Neurochem. 2005 Dec;95(6):1794-801. doi: 10.1111/j.1471-4159.2005.03511.x. Epub 2005 Oct 17. PMID 16236028
- [Background] Rakel B, Cooper N, Adams HJ, Messer BR, Frey Law LA, Dannen DR, Miller CA, Polehna AC, Ruggle RC, Vance CG, Walsh DM, Sluka KA. A new transient sham TENS device allows for investigator blinding while delivering a true placebo treatment. J Pain. 2010 Mar;11(3):230-8. doi: 10.1016/j.jpain.2009.07.007. Epub 2009 Nov 27. PMID 19945354
- [Background] Liebano RE, Rakel B, Vance CGT, Walsh DM, Sluka KA. An investigation of the development of analgesic tolerance to TENS in humans. Pain. 2011 Feb;152(2):335-342. doi: 10.1016/j.pain.2010.10.040. Epub 2010 Dec 8. PMID 21144659
- [Background] Moran F, Leonard T, Hawthorne S, Hughes CM, McCrum-Gardner E, Johnson MI, Rakel BA, Sluka KA, Walsh DM. Hypoalgesia in response to transcutaneous electrical nerve stimulation (TENS) depends on stimulation intensity. J Pain. 2011 Aug;12(8):929-35. doi: 10.1016/j.jpain.2011.02.352. Epub 2011 Apr 9. PMID 21481649
- [Background] Pantaleao MA, Laurino MF, Gallego NL, Cabral CM, Rakel B, Vance C, Sluka KA, Walsh DM, Liebano RE. Adjusting pulse amplitude during transcutaneous electrical nerve stimulation (TENS) application produces greater hypoalgesia. J Pain. 2011 May;12(5):581-90. doi: 10.1016/j.jpain.2010.11.001. Epub 2011 Feb 1. PMID 21277840
- [Background] DeSantana JM, Walsh DM, Vance C, Rakel BA, Sluka KA. Effectiveness of transcutaneous electrical nerve stimulation for treatment of hyperalgesia and pain. Curr Rheumatol Rep. 2008 Dec;10(6):492-9. doi: 10.1007/s11926-008-0080-z. PMID 19007541
- [Background] Arnold LM, Crofford LJ, Mease PJ, Burgess SM, Palmer SC, Abetz L, Martin SA. Patient perspectives on the impact of fibromyalgia. Patient Educ Couns. 2008 Oct;73(1):114-20. doi: 10.1016/j.pec.2008.06.005. Epub 2008 Jul 21. PMID 18640807
- [Background] Choy EH, Arnold LM, Clauw DJ, Crofford LJ, Glass JM, Simon LS, Martin SA, Strand CV, Williams DA, Mease PJ. Content and criterion validity of the preliminary core dataset for clinical trials in fibromyalgia syndrome. J Rheumatol. 2009 Oct;36(10):2330-4. doi: 10.3899/jrheum.090368. PMID 19820222
- [Background] Walsh DM, Howe TE, Johnson MI, Sluka KA. Transcutaneous electrical nerve stimulation for acute pain. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006142. doi: 10.1002/14651858.CD006142.pub2. PMID 19370629
- [Background] Noehren B, Dailey DL, Rakel BA, Vance CG, Zimmerman MB, Crofford LJ, Sluka KA. Effect of transcutaneous electrical nerve stimulation on pain, function, and quality of life in fibromyalgia: a double-blind randomized clinical trial. Phys Ther. 2015 Jan;95(1):129-40. doi: 10.2522/ptj.20140218. Epub 2014 Sep 11. PMID 25212518
- [Derived] Chimenti RL, Rakel BA, Dailey DL, Vance CGT, Zimmerman MB, Geasland KM, Williams JM, Crofford LJ, Sluka KA. Test-Retest Reliability and Responsiveness of PROMIS Sleep Short Forms Within an RCT in Women With Fibromyalgia. Front Pain Res (Lausanne). 2021 Jun 8;2:682072. doi: 10.3389/fpain.2021.682072. eCollection 2021. PMID 35295526
- [Derived] Vance CGT, Zimmerman MB, Dailey DL, Rakel BA, Geasland KM, Chimenti RL, Williams JM, Golchha M, Crofford LJ, Sluka KA. Reduction in movement-evoked pain and fatigue during initial 30-minute transcutaneous electrical nerve stimulation treatment predicts transcutaneous electrical nerve stimulation responders in women with fibromyalgia. Pain. 2021 May 1;162(5):1545-1555. doi: 10.1097/j.pain.0000000000002144. PMID 33230010
- [Derived] Merriwether EN, Agalave NM, Dailey DL, Rakel BA, Kolker SJ, Lenert ME, Spagnola WH, Lu Y, Geasland KM, Allen LH, Burton MD, Sluka KA. IL-5 mediates monocyte phenotype and pain outcomes in fibromyalgia. Pain. 2021 May 1;162(5):1468-1482. doi: 10.1097/j.pain.0000000000002089. PMID 33003107
- [Derived] Dailey DL, Vance CGT, Rakel BA, Zimmerman MB, Embree J, Merriwether EN, Geasland KM, Chimenti R, Williams JM, Golchha M, Crofford LJ, Sluka KA. Transcutaneous Electrical Nerve Stimulation Reduces Movement-Evoked Pain and Fatigue: A Randomized, Controlled Trial. Arthritis Rheumatol. 2020 May;72(5):824-836. doi: 10.1002/art.41170. Epub 2020 Mar 18. PMID 31738014
- [Derived] Merriwether EN, Frey-Law LA, Rakel BA, Zimmerman MB, Dailey DL, Vance CGT, Golchha M, Geasland KM, Chimenti R, Crofford LJ, Sluka KA. Physical activity is related to function and fatigue but not pain in women with fibromyalgia: baseline analyses from the Fibromyalgia Activity Study with TENS (FAST). Arthritis Res Ther. 2018 Aug 29;20(1):199. doi: 10.1186/s13075-018-1671-3. PMID 30157911
- [Derived] Dailey DL, Frey Law LA, Vance CG, Rakel BA, Merriwether EN, Darghosian L, Golchha M, Geasland KM, Spitz R, Crofford LJ, Sluka KA. Perceived function and physical performance are associated with pain and fatigue in women with fibromyalgia. Arthritis Res Ther. 2016 Mar 16;18:68. doi: 10.1186/s13075-016-0954-9. PMID 26979999
- See also: Link for Dr. Crofford — https://labnodes.vanderbilt.edu/member/profile/id/10689
- See also: Dr. Kathleen Sluka — http://www.medicine.uiowa.edu/pt/pain/
- See also: Dr. Dana Dailey and Dr. Carol Vance — https://medicine.uiowa.edu/pt/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TENS: Active TENS for 4 weeks of the study and will add an additional 4 weeks of active TENS for the last 4 weeks of the study.
  TENS: TENS Parameters: Active TENS and Placebo TENS
  * TENS Frequency - 10 to100 Hz
  * TENS Pulse Width - 200 µs
  * TENS Intensity - Maximal tolerable intensity
  * Duration: 2 hours per day. The 2 hours may be broken into smaller segments of time with a minimum of 30 minutes.
  * Administration - Daily
  * TENS Location: TENS electrode on the skin will be a 4 x 7 butterfly electrode to the cervical and lumbar region.
  Placebo TENS Unit Active TENS unit Stand Care - no TENS
- Placebo TENS: This group will receive placebo TENS for the first 4 weeks of the study and then active TENS for the last four weeks of the study.
  TENS: TENS Parameters: Active TENS and Placebo TENS
  * TENS Frequency - 10 to100 Hz
  * TENS Pulse Width - 200 µs
  * TENS Intensity - Maximal tolerable intensity
  * Duration: 2 hours per day. The 2 hours may be broken into smaller segments of time with a minimum of 30 minutes.
  * Administration - Daily
  * TENS Location: TENS electrode on the skin will be a 4 x 7 butterfly electrode to the cervical and lumbar region.
  Placebo TENS Unit Active TENS unit Stand Care - no TENS
- No TENS (Standard Care): Subjects will not receive TENS intervention during the first 4 weeks of the trial but will complete all testing procedures as the other two arms. This group will receive active TENS during the last 4 weeks of the study.
Period: Overall Study
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Started | 103 | 99 | 99
Completed (Per Protocol, completed visit 3) | 76 | 68 | 94
Not Completed | 27 | 31 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Withdrawal by Subject | 15 | 11 | 4
Not completed — Minimum dose not met | 10 | 16 | 0
Not completed — Given wrong unit (placebo) | 1 | 0 | 0
Not completed — Excluded for prior TENS | 0 | 1 | 0
Not completed — Researcher Termination of Participant | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TENS | Placebo TENS | no TENS (Standard Care) | Total
Number analyzed (Participants) | 103 | 99 | 99 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 93 | 95 | 285
  >=65 years | 6 | 6 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (14.3) | 47.2 (12.6) | 48.6 (11.8) | 46.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 99 | 99 | 301
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 15
  Not Hispanic or Latino | 96 | 92 | 88 | 276
  Unknown or Not Reported | 2 | 2 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 5 | 0 | 0 | 5
  Black or African American | 0 | 5 | 3 | 8
  White | 90 | 87 | 85 | 262
  More than one race | 4 | 3 | 5 | 12
  Unknown or Not Reported | 1 | 1 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 103 | 99 | 99 | 301
Pain with movement six minute walk test [Mean (Standard Deviation); unit: 0 to 10 low to high scale] | 6.5 (1.9) | 6.2 (1.9) | 6.4 (1.9) | 6.4 (1.9)
Pain with movement five time sit to stand [Mean (Standard Deviation); unit: 0 to 10 low to high scale] | 5.8 (2.4) | 5.5 (2.2) | 5.6 (2.2) | 5.6 (2.2)
Pain at rest [Mean (Standard Deviation); unit: 0 to 10 low to high scale] | 6.2 (1.5) | 5.9 (1.4) | 6.1 (1.6) | 6.0 (1.5)
Fatigue at rest [Mean (Standard Deviation); unit: 0 to 10 low to high scale] | 6.8 (2.0) | 6.1 (1.8) | 6.4 (2.0) | 6.43 (1.9)
Fibromyalgia Impact Questionnaire Revised - Pain [Mean (Standard Deviation); unit: 0 to 10 low to high scale] | 6.7 (1.8) | 6.0 (1.6) | 6.15 (1.8) | 6.28 (1.7)
Fibromyalgia Impact Questionnaire Revised [Mean (Standard Deviation); unit: Scoring 0 to 100 low to high scale] | 59.2 (16.8) | 53.7 (15.9) | 55.6 (16.0) | 56.1 (16.2)
Short Form 36 Physical Component Score [Median (Standard Deviation); unit: T-score mean of 50] — The SF36 Physical Functioning Component Score (PCS) quality of life measure. A T-Score of 50 represents the mean, with a standard deviation of 10, values less than 50 indicate a less than average score while values greater than 50 indicate greater than average scores" . Higher T-scores reflect better quality of life and lower T-score reflect lesser quality of life
  T-score mean of 50 | 32.7 (6.4) | 33.3 (6.2) | 32.7 (6.6) | 32.9 (6.4)
Short Form 36 Mental Health Component Score [Mean (Standard Deviation); unit: T-score mean of 50] — The SF36 Mental Health Component Scale (MCS) quality of life measure. A T-Score of 50 represents the mean, with a standard deviation of 10, values less than 50 indicate a less than average score while values greater than 50 indicate greater than average scores" . Higher T-scores reflect better quality of life and lower T-score reflect lesser quality of life
  T-score mean of 50 | 38.7 (10.0) | 40.2 (10.2) | 39.5 (10.6) | 39.4 (10.2)
Tampa Scale of Kinesiophobia [Mean (Standard Deviation); unit: Scoring 17 to 68 low to high] | 36.5 (7.7) | 37.1 (8.0) | 37.4 (8.3) | 37 (8.0)
Six minute walk test (Feet) [Mean (Standard Deviation); unit: Feet] | 1386 (323) | 1358 (305) | 1316 (318) | 1353.3 (315)
Five time sit to stand [Mean (Standard Deviation); unit: sit-to-stand repetitions/10 seconds] | 4.1 (1.5) | 4.0 (1.4) | 3.9 (1.5) | 4.0 (1.4)
Physical Activity (Moderate-Vigorous) [Mean (Full Range); unit: Average Minute/Day] | 17.7 [7.4 to 29.0] | 16.5 [6.3 to 29.1] | 15.0 [7.3 to 36.0] | 16.4 [6.3 to 36.0]

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating With Movement (0-10 Low to High Scale) During Six Minute Walk Test
Description: Numeric rating scale of 0-10 (low to high scale) for pain with movement during six minute walk test; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Units on a scale
  Change at 4 weeks | -1.8 [-2.3 to -1.2] | -0.8 [-1.4 to -0.2] | 0.00 [-0.5 to 0.6]
  Change at 8 weeks | -2.0 [-2.8 to -1.3] | -1.9 [-2.7 to -1.2] | -1.9 [-2.6 to -1.2]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2-Visit 3; Test type: Superiority; p = 0.008, Linear mixed models for repeated measure — To account for multiple tests involving pairwise treatment group comparisons, p-values were adjusted using Bonferroni's method; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.8 to -0.2]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.6 to -1.0]

2. Primary Outcome: Pain Rating With Movement (0-10 Low to High Scale) During Five Time Sit to Stand Test
Description: Numeric rating scale of 0-10 for pain with movement with five time sit to stand test. Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -1.6 [-2.30 to -1.0] | -0.3 [-1.0 to 0.3] | 0.2 [-0.4 to 0.9]
  Change at 8 weeks | -1.9 [-2.6 to -1.1] | -1.4 [-2.2 to -0.7] | -1.3 [-2.1 to -0.6]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.002, Linear mixed models for repeated measure; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.2 to -0.4]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.8 to -1.0]

3. Secondary Outcome: Resting Pain (0-10 Low to High Scale)
Description: Numeric rating scale of 0-10 for resting pain; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Baseline, Visit 2 to Visit 3 (4 weeks, randomized to 3 groups) and Visit 4 (4 weeks, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -1.9 [-2.5 to -1.4] | -0.7 [-1.3 to -0.1] | -0.5 [-1.1 to 0.00]
  Change at 8 weeks | -2.2 [-2.9 to -1.6] | -1.9 [-2.6 to -1.2] | -2.2 [-2.8 to -1.5]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.0006, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.1 to -0.4]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.2 to -0.6]

4. Secondary Outcome: Fatigue Rating (0-10 Low to High Scale) During Six Minute Walk Test
Description: Fatigue measured with 0-10 numeric rating scale during six minute walk test; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Units on a scale
  Change at 4 weeks | -1.5 [-2.2 to -0.8] | -0.1 [-0.9 to 0.7] | 0.4 [-0.3 to 1.1]
  Change at 8 weeks | -1.3 [-2.0 to -0.6] | -0.9 [-1.7 to -0.2] | -0.9 [-1.7 to -0.2]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.4 to -0.4]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -0.9]

5. Secondary Outcome: Fatigue Rating (0-10 Low to High Scale) During Five Time Sit to Stand
Description: Fatigue measured by 0-10 numeric rating scale after five time sit to stand; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Units on a scale
  Change at 4 weeks | -1.2 [-1.9 to -0.5] | -0.0 [-0.8 to 0.7] | 0.8 [0.1 to 1.5]
  Change at 8 weeks | -1.1 [-1.9 to -0.4] | -0.8 [-1.6 to -0.1] | -0.6 [-1.4 to 0.1]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.011, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.2]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.0 to -1.0]

6. Secondary Outcome: Resting Fatigue Rating (0-10 Low to High Scale)
Description: Fatigue measured at rest with a 0-10 numeric rating scale; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Population: Baseline, Visit 2 to Visit 3 (4 weeks, randomized to 3 groups) and Visit 4 (4 weeks, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Units on a scale
  Change at 4 weeks | -1.9 [-2.6 to -1.2] | -0.8 [-1.5 to -0.04] | -0.4 [-1.0 to 0.4]
  Change at 8 weeks | -2.1 [-2.9 to -1.4] | -1.6 [-2.4 to -0.8] | -1.8 [-2.6 to -1.1]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.016, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.1]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.0002, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.6 to -0.6]

7. Secondary Outcome: Fibromyalgia Impact Questionnaire Revised
Description: Disease Impact self report Questionnaire, Scoring 0-100; higher score indicates greater disease impact; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Active TENS: Active TENS for 4 weeks of the study and will add an additional 4 weeks of active TENS for the last 4 weeks of the study.
  TENS: TENS Parameters: Active TENS and Placebo TENS
  * TENS Frequency - 2-125 Hz
  * TENS Pulse Width - 200 µs
  * TENS Intensity - Maximal tolerable intensity
  * Duration: 2 hours per day. The 2 hours may be broken into smaller segments of time with a minimum of 30 minutes.
  * Administration - Daily
  * TENS Location: TENS electrode on the skin will be a 4 x 7 butterfly electrode to the cervical and lumbar region.
  Placebo TENS Unit Active TENS unit Stand Care - no TENS
- Placebo TENS: This group will receive placebo TENS for the first 4 weeks of the study and then active TENS for the last four weeks of the study.
  TENS: TENS Parameters: Active TENS and Placebo TENS
  * TENS Frequency - 2-125 Hz
  * TENS Pulse Width - 200 µs
  * TENS Intensity - Maximal tolerable intensity
  * Duration: 2 hours per day. The 2 hours may be broken into smaller segments of time with a minimum of 30 minutes.
  * Administration - Daily
  * TENS Location: TENS electrode on the skin will be a 4 x 7 butterfly electrode to the cervical and lumbar region.
  Placebo TENS Unit Active TENS unit Stand Care - no TENS
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Units on a scale
  Change at 4 weeks | -8.5 [-12.9 to 4.0] | -3.4 [-6.5 to 0.3] | -1.39 [-4.4 to 1.6]
  Change at 8 weeks | -9.6 [-13.8 to 5.4] | -11.1 [-15.2 to 7.0] | -10.7 [-14.8 to -6.6]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.074, Linear mixed models for repeated measure; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-10.4 to 0.3]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.005, Linear mixed models for repeated measure; Mean Difference (Final Values) = -7.1, 95% CI 2-sided [-12.4 to -1.8]

8. Secondary Outcome: Fibromyalgia Impact Questionnaire Revised - Pain Rating (0-10 Low to High Scale)
Description: numeric rating scale 0 to 10 from the Fibromyalgia Impact Questionnaire Revised: Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -1.3 [-1.8 to -0.7] | -0.4 [-0.9 to -0.2] | -0.1 [-0.6 to 0.4]
  Change at 8 weeks | -1.4 [-2.0 to -0.8] | -1.2 [-1.7 to -0.6] | -1.4 [-1.9 to -0.8]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.018, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to -0.1]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.0006, Linear mixed models for repeated measure; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.9 to -0.4]

9. Secondary Outcome: Brief Pain Inventory - Interference (0-10 Low to High Scale)
Description: Brief Pain Inventory - Interference; Score 0-10 with higher score indicating greater interference; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -0.9 [-1.4 to -0.5] | -0.3 [-0.7 to 0.2] | -0.3 [-0.7 to 0.2]
  Change at 8 weeks | -1.1 [-1.6 to -0.6] | -0.9 [-1.4 to -0.3] | -1.2 [-1.7 to -0.7]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.043, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to -0.01]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.048, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.3 to -0.0]

10. Secondary Outcome: Brief Pain Inventory, Intensity (0-10 Low to High Scale)
Description: Brief Pain Inventory - Interference, Scale of 0-10 with higher score indicating greater intensity; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -0.8 [-1.1 to -0.4] | -0.3 [-0.6 to 0.1] | 0.15 [-0.2 to 0.5]
  Change at 8 weeks | -1.0 [-1.4 to -0.6] | -0.9 [-1.3 to -0.5] | -0.9 [-1.2 to -0.5]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.036, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to -0.0]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p < 0.0001, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.4 to -0.4]

11. Secondary Outcome: Tampa Scale of Kinesiophobia (17 to 68 Low to High)
Description: Self report questionnaire with higher scores indicating greater kinesiophobia, score 17-68; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
units on a scale
  Change at 4 weeks | -0.7 [-2.0 to 0.6] | -0.3 [-1.7 to 1.0] | -0.2 [-1.4 to 1.1]
  Change at 8 weeks | -0.3 [-1.6 to 1.1] | -2.3 [-3.7 to -0.9] | -3.3 [-4.6 to -2.0]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.3 to 1.5]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.4 to 1.3]

12. Secondary Outcome: Short Form Survey 36; Mental Component Score (T Score Mean of 50)
Description: Multidimensional Self Report Questionnaire, T-score; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
  The SF36 Mental Health Component Score (MCS) quality of life measure. A T-Score of 50 represents the mean, with a standard deviation of 10, values less than 50 indicate a less than average score while values greater than 50 indicate greater than average scores" . Higher T-scores reflect better quality of life and lower T-score reflect lesser quality of life
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
T-Score
  Change at 4 weeks | 2.3 [0.2 to 4.4] | 1.2 [-0.9 to 3.4] | -0.04 [-2.1 to 2.0]
  Change at 8 weeks | 2.1 [-0.2 to 4.4] | 3.6 [1.3 to 6.0] | 2.8 [0.6 to 5.0]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-1.9 to 4.1]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Test type: Superiority; p = 0.17, Linear mixed models for repeated measure; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-0.6 to 5.3]

13. Secondary Outcome: Short Form Survey 36 Physical Component Score (T-score Mean of 50) Higher Scores Indicating Better Health
Description: Multidimensional self report scale, T score change; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
  The SF36 Physical Functioning Component Score (PCS) quality of life measure. A T-Score of 50 represents the mean, with a standard deviation of 10, values less than 50 indicate a less than average score while values greater than 50 indicate greater than average scores" . Higher T-scores reflect better quality of life and lower T-score reflect lesser quality of life .
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
T-Score
  Change at 4 weeks | 2.4 [1.0 to 3.7] | 1.2 [-0.2 to 2.5] | 1.4 [0.1 to 2.6]
  Change at 8 weeks | 3.5 [2.0 to 5.1] | 3.2 [1.6 to 4.8] | 4.4 [2.9 to 5.9]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.36, Linear mixed models for repeated measure; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.7 to 3.1]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.58, Linear mixed models for repeated measure; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.8 to 2.8]

14. Secondary Outcome: Six Minute Walk Test
Description: 6MWT - Feet walked as fast as comfortable in six minute; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Feet
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Feet
  Change at 4 weeks | -1 [-55 to 54] | -20 [-75 to 36] | -42.1 [-95 to 11]
  Change at 8 weeks | 15 [-42 to 71] | 16 [-41 to 74] | -2 [-57 to 53]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure; Mean Difference (Final Values) = 19, 95% CI 2-sided [-58 to 96]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure; Mean Difference (Final Values) = 42, 95% CI 2-sided [-34 to 117]

15. Secondary Outcome: Five Time Sit to Stand Test Rate Per 10 Seconds
Description: Time for sit to stand for 5 repetitions converted to a rate of number of sit to stand per 10 seconds; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: sit-to-stand repetitions/10 seconds
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
sit-to-stand repetitions/10 seconds
  Change at 4 weeks | 0.6 [0.3 to 1.0] | 0.4 [0.0 to 0.7] | 0.1 [-0.3 to 0.4]
  Change at 8 weeks | 0.6 [0.2 to 1.0] | 0.8 [0.4 to 1.3] | 0.6 [0.1 to 1.0]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p = 0.96, Linear mixed models for repeated measure; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p = 0.008, Linear mixed models for repeated measure; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.1 to 1.0]

16. Secondary Outcome: Moderate Vigorous Physical Activity Minutes Per Day
Description: Accelerometry data classification of physical activity in minutes per day, percent change; Intention to treat analysis corrected for site (Iowa and Vanderbilt) differences. Mean change (from baseline, Visit 2) at Visit 3 (after 4 weeks of home TENS use, or placebo TENS, or no TENS) and at Visit 4 (after 4 weeks of home TENS all groups) with 95% adjusted confidence intervals. Change scores are presented for the randomized phase between Visit-2 and Visit-3, and for the difference from baseline at Visit 4 when all subjects received active-TENS. p-values represent post hoc comparisons between groups
Time Frame: Time Frame: Baseline (Visit 2), 4 weeks (Visit 3, randomized to 3 groups), and 8 weeks (Visit 4, all groups home TENS)
Measure: Mean (95% Confidence Interval); unit: Minutes per day
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care)
Number analyzed (Participants) | 103 | 99 | 99
Minutes per day
  Change at 4 weeks | -9.4 [-27.8 to 13.5] | 2.5 [-18.6 to 29.1] | -14.1 [-29.5 to 4.7]
  Change at 8 weeks | -6.8 [-27.2 to 19.3] | -0.3 [-22.3 to 27.9] | -17.0 [-33.9 to 4.1]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure
Statistical Analysis 2: Comparison: Active TENS vs No TENS (Standard Care); Visit 2 to Visit 3; Test type: Superiority; p > 0.99, Linear mixed models for repeated measure

ADVERSE EVENTS:
Time Frame: Visit 1 to Visit 4, 9 weeks
Groups:
- Pre-Randomization: Participants who attended visit 1 or 2 prior to randomization to intervention
Arm/Group | Active TENS | Placebo TENS | No TENS (Standard Care) | Pre-Randomization
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/99 | 0/99 | 0/352
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/99 | 2/99 | 1/352
Other Adverse Events (participants affected / at risk) | 12/103 | 10/99 | 15/99 | 0/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=103) | Placebo TENS (N=99) | No TENS (Standard Care) (N=99) | Pre-Randomization (N=352)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject with chest pain between visits with emergency department visit and hospitalization; non-study related, recovered with treatment
Dehydration and gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant admitted to hospital for complaint of dehydration
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for depression
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=103) | Placebo TENS (N=99) | No TENS (Standard Care) (N=99) | Pre-Randomization (N=352)
Pain with testing (Nervous system disorders) | 12 (12) | 10 (10) | 15 (15) | 0 (0) — Increase in pain with testing at clinic visit
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 3 (3) | 0 (0) — Report of upper respiratory infection or difficulty during the study
Pain with TENS; At home, unspecified (General disorders) | 4 (4) | 4 (4) | 3 (3) | 0 (0)
Skin Irritation from actigraph band (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Skin Irritation with Electrodes (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Bladder Infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Sinus Infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 3 (3) | 0 (0)
Fall (General disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
Headache or Migraine (General disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Dental Procedures (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT01888640/Prot_SAP_000.pdf